CLINICAL TRIAL: NCT00119574
Title: Evaluating a Collaborative Care Model for the Treatment of Schizophrenia (EQUIP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other); asd (Unknown)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CPI 99-383; RCD 00-033; NIMH MH-5423; NIMH MH-068639
Record Dates: First submitted 2005-07-01; First posted 2005-07-13 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-07

CONDITIONS: Schizophrenia Disorders; Chronic Illness; Schizoaffective Disorder; Weight Gain
Keywords: Randomized Controlled Trial; Quality of Health Care; Health Services Research; Guidelines; Medical Informatics Computing; Services, Mental Health; Medicine, Evidence-Based; Quality Assurance, Healthcare; Quality Indicators, Health Care; Veterans
MeSH Terms: conditions — Schizophrenia; Chronic Disease; Psychotic Disorders; Weight Gain; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Collaborative Chronic Illness Model

INTERVENTIONS:
Procedure: Collaborative Chronic Illness Model

SUMMARY:
Policy makers and consumers are increasingly concerned about the quality and efficiency of care provided to individuals with severe, chronic illnesses such as schizophrenia. These illnesses are expensive to treat and present significant challenges to organizations that are responsible for providing effective care. Occurring in 1% of the United States population, schizophrenia accounts for 10% of permanently disabled people, and 2.5% of all healthcare expenditures. Clinical practice guidelines have been promulgated. Schizophrenia is treatable and outcomes can be substantially improved with the appropriate use of antipsychotic medication, caregiver education and counseling, vocational rehabilitation, and assertive treatment. However, in the VA and other mental health systems, many patients with schizophrenia receive substandard care. Methods are needed that improve the quality of usual care for this disorder while being feasible to implement at typical clinics.

To date, most efforts to improve care for schizophrenia have focused on educating clinicians or changing the financing of care, and have had limited success. We believe a more fundamental approach should be tried. While there are many potential strategies, experience in chronic medical illness and mental health support the efficacy of specific approaches. Collaborative care models are one such approach. They are a blueprint for reorganizing practice, and involve changes in division of labor and responsibility, adoption of new care protocols, and increased attention to patients' needs. Although collaborative care models have been successful in other chronic medical conditions, they have not yet been studied in the treatment of schizophrenia.

We have developed a collaborative care model for schizophrenia that builds on work in other disorders, and includes service delivery approaches that are known to be effective in schizophrenia. The model focuses on improving treatment through assertive care management, caregiver education and support, and standardized patient assessment with feedback of information to psychiatrists. This project, "EQUIP" (Enhancing Quality Utilization In Psychosis) is implementing collaborative care and evaluating its effectiveness in schizophrenia.

DETAILED DESCRIPTION:
Background:

Policy makers and consumers are increasingly concerned about the quality and efficiency of care provided to individuals with severe, chronic illnesses such as schizophrenia. These illnesses are expensive to treat and present significant challenges to organizations that are responsible for providing effective care. Occurring in 1% of the United States population, schizophrenia accounts for 10% of permanently disabled people, and 2.5% of all healthcare expenditures. Clinical practice guidelines have been promulgated. Schizophrenia is treatable and outcomes can be substantially improved with the appropriate use of antipsychotic medication, caregiver education and counseling, vocational rehabilitation, and assertive treatment. However, in the VA and other mental health systems, many patients with schizophrenia receive substandard care. Methods are needed that improve the quality of usual care for this disorder while being feasible to implement at typical clinics.

To date, most efforts to improve care for schizophrenia have focused on educating clinicians or changing the financing of care, and have had limited success. We believe a more fundamental approach should be tried. While there are many potential strategies, experience in chronic medical illness and mental health support the efficacy of specific approaches. Collaborative care models are one such approach. They are a blueprint for reorganizing practice, and involve changes in division of labor and responsibility, adoption of new care protocols, and increased attention to patients' needs. Although collaborative care models have been successful in other chronic medical conditions, they have not yet been studied in the treatment of schizophrenia.

We have developed a collaborative care model for schizophrenia that builds on work in other disorders, and includes service delivery approaches that are known to be effective in schizophrenia. The model focuses on improving treatment through assertive care management, caregiver education and support, and standardized patient assessment with feedback of information to psychiatrists. This project, "EQUIP" (Enhancing Quality Utilization In Psychosis) is implementing collaborative care and evaluating its effectiveness in schizophrenia.

Objectives:

The objective of this project was to implement the care model at two large VA mental health centers, and evaluate its effect on clinicians, the organization of care, and treatment appropriateness, utilization and outcomes in veterans with schizophrenia. We hypothesized that this care model would increase provider adherence to treatment guidelines and improve the quality of care. We planned to describe implementation of the model, and barriers and facilitators to its implementation. We planned to evaluate the model by comparing treatment under the care model with usual care. Changes in the structure of care were evaluated using qualitative methods.

Methods:

EQUIP was a controlled trial of the care model. At two VA medical centers, clinicians (n=66) and their patients (n=398) were randomized to an intervention or a control condition. In the intervention group, a chronic care model was implemented for 15 months. Before, during, and after implementation, surveys and semi-structured interviews were conducted with clinicians and managers to assess their clinical practices, competencies, expectations, experiences, and observations concerning the implementation. Data sources included patient interviews, clinician interviews, and data from VistA. The feasibility of more broadly implementing the collaborative care model was assessed utilizing qualitative and quantitative information about the model's strengths and weaknesses, factors that facilitated/impeded implementation, direct costs of implementation and maintenance, and effects on treatment service utilization.

Status:

Data collection is complete. Data analyses are ongoing. Reports are being written and published. Presentations are being given.

ELIGIBILITY:
Inclusion Criteria:

Providers (Psychiatrists, Case Managers, Nurses):

Working at one of the participating VA Mental Health Clinics

Providers: 68 Patients: 375

Patients:

* At least 18 years old
* Diagnosis of Schizophrenia, Schizoaffective, or schizophreniform disorder
* At least 2 treatment visits with a psychiatrist at the clinic during the previous 6 months.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Estimated)
Dates: Start 2002-01; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
At 15 mo.: Provider attitudes on controlling symptoms & side-effects, & on family involvement Patient clinical outcomes Throughout the study: Patient compliance Provider practice patterns & adherence to VA guidelines Patient utilization

SECONDARY OUTCOMES:
Process assessment throughout the course of the study of barriers and facilitators to the intervention�s implementation

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stehle Young, MD MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

REFERENCES:
- [Result] Niv N, Cohen AN, Sullivan G, Young AS. The MIRECC version of the Global Assessment of Functioning scale: reliability and validity. Psychiatr Serv. 2007 Apr;58(4):529-35. doi: 10.1176/ps.2007.58.4.529. PMID 17412856
- [Result] Niv N, Cohen AN, Mintz J, Ventura J, Young AS. The validity of using patient self-report to assess psychotic symptoms in schizophrenia. Schizophr Res. 2007 Feb;90(1-3):245-50. doi: 10.1016/j.schres.2006.11.011. Epub 2007 Jan 3. PMID 17204397
- [Result] Glynn SM, Cohen AN, Niv N. New challenges in family interventions for schizophrenia. Expert Rev Neurother. 2007 Jan;7(1):33-43. doi: 10.1586/14737175.7.1.33. PMID 17187495
- [Result] Erhart SM, Young AS, Marder SR, Mintz J. Clinical utility of magnetic resonance imaging radiographs for suspected organic syndromes in adult psychiatry. J Clin Psychiatry. 2005 Aug;66(8):968-73. doi: 10.4088/jcp.v66n0802. PMID 16086610
- [Result] Young AS, Mintz J, Cohen AN, Chinman MJ. A network-based system to improve care for schizophrenia: the Medical Informatics Network Tool (MINT). J Am Med Inform Assoc. 2004 Sep-Oct;11(5):358-67. doi: 10.1197/jamia.M1492. Epub 2004 Jun 7. PMID 15187072
- [Result] Young AS, Mintz J, Cohen AN. Using information systems to improve care for persons with schizophrenia. Psychiatr Serv. 2004 Mar;55(3):253-5. doi: 10.1176/appi.ps.55.3.253. No abstract available. PMID 15001724
- See also: Tour of the Medical Informatics Tool (MINT) which was developed and utilized to support the intervention — http://www.npistat.com/mint-tour